CLINICAL TRIAL: NCT03607058
Title: Ataksik Hastalarda Oyun Temelli Egzersiz Eğitiminin Denge ve Postural Kontrol Üzerine Etkisi
Brief Title: The Effects of Game Based Exercise Training on Balance and Postural Control in Patients With Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ÖZGE ONURSAL KILINÇ, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KA-17049
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Ataxia
MeSH Terms: conditions — Ataxia | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect + Exercise Training (Active Comparator): Xbox Kinect and exercise training will be applied together for 8 weeks. Selected balance, coordination and walking exercises according to the individual needs of patients. A treatment session in this arm will consist of Kinect games for 40 minutes and exercise training for 20 minutes. In this arm, patients will play each game as two repetitions. Each game lasts about 3-4 minutes, and patients will be seated for resting between the games. After 10 weeks washout period only exercise training will be applied for 8 weeks.
  Interventions: Other: Kinect + Exercise Training
- Exercise Training (Active Comparator): Exercise training will be applied for 8 weeks. Selected balance, coordination and walking exercises according to the individual needs of patients. After 10 weeks washout period exercise training and Xbox Kinect will be applied together for 8 weeks.
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Kinect + Exercise Training — Kinect + Exercise Training : Patients will play Xbox Kinect games for 40 minutes and take the treatment for 20 minutes, 3 days in a week for 8 weeks. After 10 weeks washout period, patients will take the treatment 1-hour, 3 days in a week for 8 weeks.
  Arms: Kinect + Exercise Training
Other: Exercise Training — Exercise Training: Patients will take the treatment 1-hour, 3 days in a week for 8 weeks. After 10 weeks washout period, patients will play Xbox Kinect games for 40 minutes and take the treatment for 20 minutes, 3 days in a week for 8 weeks.
  Arms: Exercise Training

SUMMARY:
This study was planned to investigate the effects of exercise training based on Microsoft Kinect application on balance and postural control in ataxic patients.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be divided into two groups randomly: 'Kinect and exercise training' and 'exercise training'. The assessments will be made by a blind investigator four times, before and after the implementation of both protocols. The evaluations will take approximately 1 hour. The demographic information of the cases will be recorded. Designed as cross over study, two treatment protocols will be used in this study. The first protocol will be Xbox Kinect application plus exercise program, the second protocol will be only exercise program. At the beginning of the study, 2 groups will be allocated (Group A and Group B) randomly. For group A, the Xbox Kinect application plus exercise program will be applied for the first 8 weeks. For group B, only exercise program will be applied therapy first 8 weeks. All assessments will be repeated before and after each therapy period. Exercise program will consist of selected balance, coordination and walking exercises according to the individual needs of patients. After 10 weeks washout period, patients will be included in the other group. All patients will take the treatment 1-hour, 3 days in a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ataxia
* Ataxic patients who are able to walk 25 m independently
* Ataxic patients who had a Mini Mental Test Score of 24 points and over;

Exclusion Criteria:

* Clinical diagnosis of systemic problems (Diabetes Mellitus, Hypertension)
* Clinical diagnosis of cognitive impairment
* Patients who have fallen at least once in the last 6 months
* Patients who had Berg Balance Scale score of 40 points and below

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Limits of Stability Test of Neurocom Balance Master (Static Posturography) | change from baseline in dynamic balance component of postural control at 8 weeks
  Limits of stability test (LOS) assesses dynamic balance during the performance of specific tasks with visual feedback. It quantifies objectively the maximum distance a person can lean in a given direction without losing balance, stepping or reaching for assistance

SECONDARY OUTCOMES:
International Cooperative Ataxia Rating Scale | change from baseline in severity of ataxic symptoms at 8 weeks
  The International Cooperative Ataxia Rating Scale was developed to quantify the level of impairment as a result of ataxia as related to hereditary ataxias. The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. the maximum score is 100, the minimum score is 0 in this scale. Higher scores indicate higher levels of impairment. Postural and gait disturbances subscale has 7 items (0-34 points), limb ataxia subscale has 7 items (0-52 points), Dysarthria subscale has 2 items (0-4 points) and oculomotor disorders subscale has 3 items (0-6 points). The total score is obtained by summing the scores of the sub-scales.
Timed Up and Go test (TUG) | change from baseline in falling risk at 8 weeks
  TUG was developed to determine falling risk and measure the progress of balance, sit to stand, and walking.
Functional Reach Test (FRT) | change from baseline in dynamic balance at 8 weeks
  FRT is a quick and simple, single-task dynamic test that defines functional reach as "the maximal distance one can reach forward beyond arm's length, while maintaining a fixed base of support in the standing position". It is a dynamic rather than a static test and measures a person's "margin of stability" as well as ability to maintain balance during a functional task.
10 meter Walk Test (10mWT) | change from baseline in gait speed at 8 weeks
  The 10mWTis a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility and gait.
Trunk Impairment Scale | change from baseline in impairment of trunk at 8 weeks
  It was developed to measure the motor impairment of the trunk through the evaluation of static and dynamic sitting balance as well as co-ordination of trunk movement. Three subscales: static sitting balance, dynamic sitting balance and coordination. There are 17 items in this scale and for each item, a 2-, 3- or 4-point ordinal scale is used. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. The total score for this scale ranges between 0 for a minimal performance to 23 for a perfect performance. The total score is obtained by summing the scores of the subscales.
Dynamic Gait Index (DGI) | change from baseline in balance, fall risk and gait at 8 weeks
  The DGI was developed as a clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks. The DGI was developed as a clinical tool to assess gait, balance and fall risk. It evaluates not only usual steady-state walking, but also walking during more challenging tasks. 8 functional walking tests are performed by the subject and marked out of three according to the lowest category which applies. 24 is the total individual score possible. Scores of 19 or less have been related to increase incidence of falls.
Berg Balance Scale (BBS) | change from baseline in balance performance at 8 weeks
  A 14-item objective measure designed to assess static balance and fall risk. Static and dynamic activities of varying difficulty are performed.Item-level scores range from 0-4, determined by ability to perform the assessed activity. Item scores are summed. Maximum score is 56.
Rhythmic Weight Shift (RWS) of Neurocom Balance Master (Static Posturography) | change from baseline in directional control and movement velocity while move the center of gravity at 8 weeks
  RWS test quantifies the patient's ability to rhythmically move their Center of Gravity (COG) from left to right (lateral) and forward to backward (anterior/ posterior) between two targets at three distinct speeds: slow, medium, and fast.
Unilateral Stance Test (US) of Neurocom Balance Master (Static Posturography) | change from baseline in postural sway velocity at 8 weeks
  The US quantifies postural sway velocity with the patient standing on either the right or left foot with eyes open and with eyes closed.
Weight Bearing Squat (WBS) of Neurocom Balance Master (Static Posturography) | change from baseline in weight bearing at 8 weeks
  During the WBS, the patient is instructed to maintain equal weight on each leg while standing erect and then squatting in three positions of knee flexion. The percentage of body weight borne by each leg is measured with the patient standing at 0° (erect), 30°, 60°, and 90° of knee flexion.
Walk Across (WA) of Neurocom Balance Master (Static Posturography) | change from baseline in gait characteristics at 8 weeks
  The WA quantifies characteristics of gait as the patient walks across the length of the force plate. The test characterizes steady state gait by having the patient begin well behind and continuing beyond the force plate. Measured parameters are average step width, average step length, speed and step length symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Özge ONURSAL KILINÇ, Msc, Principal Investigator — Hacettepe University; Ender AYVAT, PhD, Principal Investigator — Hacettepe University; Fatma AYVAT, Msc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yelnik A, Bonan I. Clinical tools for assessing balance disorders. Neurophysiol Clin. 2008 Dec;38(6):439-45. doi: 10.1016/j.neucli.2008.09.008. Epub 2008 Oct 18. PMID 19026963
- [Result] Trouillas P, Takayanagi T, Hallett M, Currier RD, Subramony SH, Wessel K, Bryer A, Diener HC, Massaquoi S, Gomez CM, Coutinho P, Ben Hamida M, Campanella G, Filla A, Schut L, Timann D, Honnorat J, Nighoghossian N, Manyam B. International Cooperative Ataxia Rating Scale for pharmacological assessment of the cerebellar syndrome. The Ataxia Neuropharmacology Committee of the World Federation of Neurology. J Neurol Sci. 1997 Feb 12;145(2):205-11. doi: 10.1016/s0022-510x(96)00231-6. PMID 9094050
- [Result] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Result] Berg KO, Maki BE, Williams JI, Holliday PJ, Wood-Dauphinee SL. Clinical and laboratory measures of postural balance in an elderly population. Arch Phys Med Rehabil. 1992 Nov;73(11):1073-80. PMID 1444775
- [Result] Lange B, Chang CY, Suma E, Newman B, Rizzo AS, Bolas M. Development and evaluation of low cost game-based balance rehabilitation tool using the Microsoft Kinect sensor. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:1831-4. doi: 10.1109/IEMBS.2011.6090521. PMID 22254685
- [Result] Donath L, Rossler R, Faude O. Effects of Virtual Reality Training (Exergaming) Compared to Alternative Exercise Training and Passive Control on Standing Balance and Functional Mobility in Healthy Community-Dwelling Seniors: A Meta-Analytical Review. Sports Med. 2016 Sep;46(9):1293-309. doi: 10.1007/s40279-016-0485-1. PMID 26886474
- [Result] Shih MC, Wang RY, Cheng SJ, Yang YR. Effects of a balance-based exergaming intervention using the Kinect sensor on posture stability in individuals with Parkinson's disease: a single-blinded randomized controlled trial. J Neuroeng Rehabil. 2016 Aug 27;13(1):78. doi: 10.1186/s12984-016-0185-y. PMID 27568011
- [Result] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Result] Peters DM, Fritz SL, Krotish DE. Assessing the reliability and validity of a shorter walk test compared with the 10-Meter Walk Test for measurements of gait speed in healthy, older adults. J Geriatr Phys Ther. 2013 Jan-Mar;36(1):24-30. doi: 10.1519/JPT.0b013e318248e20d. PMID 22415358
- [Derived] Ayvat E, Onursal Kilinc O, Ayvat F, Savcun Demirci C, Aksu Yildirim S, Kursun O, Kilinc M. The Effects of Exergame on Postural Control in Individuals with Ataxia: a Rater-Blinded, Randomized Controlled, Cross-over Study. Cerebellum. 2022 Feb;21(1):64-72. doi: 10.1007/s12311-021-01277-0. Epub 2021 May 11. PMID 33973141